CLINICAL TRIAL: NCT07350187
Title: Prospective, Randomized, Controlled Trial Comparing Self-Gripping and Conventional Mesh in Laparoscopic Totally Extra Peritoneal Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TEP001
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2024-10

CONDITIONS: Inguinal Hernias
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Self-gripping mesh (Progrip™) (Experimental): Participants assigned to this arm undergo laparoscopic totally extraperitoneal (TEP) inguinal hernia repair using a self-gripping mesh (Progrip™). The mesh is positioned in the preperitoneal space without the use of additional fixation devices, relying on its microgrip technology for adherence. All other aspects of the surgical procedure are standardized.
  Interventions: Device: Self-gripping mesh (Progrip™)
- Conventional mesh with tacker fixation (Parietex™) (Active Comparator): Participants assigned to this arm undergo laparoscopic totally extraperitoneal (TEP) inguinal hernia repair using a conventional mesh (Parietex™). The mesh is fixed with a single permanent tacker placed on the pubic bone to ensure mesh stability. No fixation is applied to muscle or nerve-bearing areas. All other aspects of the surgical procedure are standardized.
  Interventions: Device: Conventional mesh with tacker fixation (Parietex™)

INTERVENTIONS:
Device: Self-gripping mesh (Progrip™) — self-gripping surgical mesh used during laparoscopic totally extraperitoneal (TEP) inguinal hernia repair. The mesh adheres to surrounding tissue via resorbable microgrips and does not require additional fixation devices.
  Arms: Self-gripping mesh (Progrip™)
Device: Conventional mesh with tacker fixation (Parietex™) — A conventional surgical mesh used during laparoscopic totally extraperitoneal (TEP) inguinal hernia repair. The mesh is fixed with a single permanent tacker placed on the pubic bone to ensure mesh stability.
  Arms: Conventional mesh with tacker fixation (Parietex™)

SUMMARY:
This study is a single-center, prospective, randomized controlled trial designed to compare clinical outcomes between self-gripping mesh and conventional mesh with limited tacker fixation in laparoscopic totally extraperitoneal (TEP) inguinal hernia repair.

Adult patients diagnosed with inguinal hernia and scheduled for laparoscopic TEP repair are randomly assigned to receive either a self-gripping mesh (Progrip™) or a conventional mesh fixed with a single permanent tacker to the pubic bone (Parietex™). Both meshes are commonly used in clinical practice and approved for inguinal hernia repair.

The primary objective of this study is to evaluate postoperative discomfort and quality of life following surgery. Outcomes are assessed using validated patient-reported questionnaires, including the Carolina Comfort Scale (CCS) and the International Prostate Symptom Score (IPSS). Secondary outcomes include postoperative complications, physical examination findings such as local induration or tenderness, operative time, and short-term hernia recurrence.

Patients are followed at 1 week, 3 weeks, and 3 months after surgery. The results of this study aim to provide comparative evidence regarding the safety and short-term clinical outcomes of self-gripping versus tacker-fixed conventional mesh in laparoscopic TEP inguinal hernia repair.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 19 to 100 years Diagnosed with inguinal hernia Scheduled to undergo laparoscopic totally extraperitoneal (TEP) inguinal hernia repair Able to understand the study procedures and provide written informed consent

Exclusion Criteria:

Patients receiving immunosuppressive therapy or with immune-related diseases Patients with urological conditions requiring urinary catheterization preoperatively or intraoperatively Patients with complicated inguinal hernia, including irreducible hernia or hernia associated with bowel injury Patients with unintended intraoperative injury during surgery Pregnant women or women of childbearing potential without confirmed non-pregnant status Patients who decline to participate or withdraw informed consent

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Postoperative discomfort assessed by the Carolina Comfort Scale (CCS) | From baseline to 1 week and 3 months after surgery
  Postoperative discomfort and quality of life are assessed using the Carolina Comfort Scale (CCS), a validated hernia-specific questionnaire evaluating pain, mesh sensation, and limitation of movement during daily activities.

SECONDARY OUTCOMES:
Postoperative urinary symptoms assessed by the International Prostate Symptom Score (IPSS) | From baseline to 1 week and 3 months after surgery
  Lower urinary tract symptoms are evaluated using the International Prostate Symptom Score (IPSS), a validated patient-reported questionnaire.
Incidence of postoperative complications | Up to 3 months after surgery
  Postoperative complications including seroma, hematoma, urinary retention, wound-related complications, and hernia recurrence are recorded.
Postoperative physical examination findings | 1 week and 3 months after surgery
  Physical examination findings such as local induration, tenderness, and abdominal wall stiffness at the surgical site are assessed during follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No